CLINICAL TRIAL: NCT02578212
Title: Trust Game and Placebo Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EKNZ 2014-396
Record Dates: First submitted 2015-10-12; First posted 2015-10-16 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Placebo Effect; Pain; Trust
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): All participants will also be introduced to the control cream: "This cream is a control cream".
  Interventions: Other: Placebo
- Placebo (Sham Comparator): All participants will then be introduced to an analgesia expectation: "This cream is a powerful pain killer", while receiving an inert cream. In this study participants will be told that they will receive a potent painkiller as well as a control cream. Making use of placebo cream is an established method to induce placebo expectations . Moreover, to increase the analgesic effect, heat pain stimuli intensity will be surreptitiously lowered for the placebo trials to a temperature corresponding to 30% of the VAS intensity and to 60% for the control trials. As the occurrence of a placebo response is highly dependent on expectations, the deceptive procedure described above is used in order to maximally enhance expectations and therefore placebo response. Participants will be debriefed after the completion of study participation.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo

SUMMARY:
In the proposed study, investigators aim to investigate the role of interpersonal trust in the conditioned placebo analgesia process with healthy male subjects in a standardized experimental heat pain paradigm.

ELIGIBILITY:
Inclusion Criteria:

* Men: age between 18 and 40 years old
* Healthy by self-report statement, thus no known current or chronic somatic diseases or psychiatric disorders
* Right-handedness (Oldfield, 1971)
* Willing to participate in study

Exclusion Criteria:

* Any acute or chronic disease (chronic pain, hypertension, heart disease, renal disease, liver disease, diabetes) as well as skin pathologies, neuropathies or nerve entrapment symptoms, sensory abnormalities affecting the tactile or thermal modality
* Current medications (psychoactive medication, narcotics, intake of analgesics) or being currently in psychological or psychiatric treatment
* Insufficient German language skills to understand the instructions
* Previous participation in studies using pain assessment (threshold and tolerance) with Peltier Devices
* Daily consumption of more than three alcoholic standard beverages per day (a standard alcoholic beverage is defined as either 3dl beer or 1 dl wine or 2cl spirits
* Current or regular drug consumption (THC, cocaine, heroin, etc.)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) rating (Intensity + unpleasantness of pain) | 2 hours

SECONDARY OUTCOMES:
Visual analogue scale (VAS) rating (trust) | 2 hours
State-Trait-Anxiety (STAI- X1) | 2 hours
State Trait Anger Expression (STAXI) | 2 hours
Questionnaire about expectations (Erwartungsfragebogen) | 2 hours
Questionnaire about the investigator (Fragebogen zum Versuchsleiter | 2 hours
sociodemographic questionnaire (Soziodemographischer Fragebogen (SES)) | 2 hours
Questionnaire about Self-assessment of partnership binding (Bochumer Bindungsfragebogen - BoBi) | 2 hours
State-Trait-Anxiety (STAI-X2 ) | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jens Gaab, Prof, Study Chair — Clinical Psychology and Psychotherapy, Department of Psychology, University of Basel
Locations (1):
- University of Basel, Basel, Switzerland